CLINICAL TRIAL: NCT00955552
Title: A Multi-center, Randomized, Double Blind, Comparative of Efficacy and Safety From Association of Capsules Glucosamine and Chondroitin Sulfate (Eurofarma) Versus Cosamin DS to Treatment With Osteoarthrosis of the Knee
Brief Title: Efficacy and Safety Study of Glucosamine/Chondroitin Sulfate to Patients Treatment With Osteoarthrosis of the Knee
Acronym: Artico
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EF-093
Record Dates: First submitted 2009-08-05; First posted 2009-08-10 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis (OA); knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Glucosamine; Chondroitin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cosamin DS® (Active Comparator): glucosamine hydrochloride 500 mg and chondroitin sulfate 400 mg (Cosamin DS®, Nutramax Laboratories).
  The medication was supplied as capsules, with the daily dose of 3 capsules.
  Interventions: Drug: Cosamin DS® (Nutramax)
- Glucosamine/ chondroitin sulphate (Experimental): Glucosamine hydrochloride 500 mg and chondroitin sulphate 400 mg association (Eurofarma) T.I.D. before each meal The medication was supplied as capsules, with the daily dose of 3 capsules.
  Interventions: Drug: Glucosamine sulphate and chondroitin sulphate association

INTERVENTIONS:
Drug: Glucosamine sulphate and chondroitin sulphate association — glucosamine sulphate 500 mg and chondroitin sulphate 400 mg association T.I.D. before each meal
  Other Names: Glucosamine sulphate and Chondroitin sulphate
  Arms: Glucosamine/ chondroitin sulphate
Drug: Cosamin DS® (Nutramax) — oral capsule of glucosamine hydrochloride 500 mg + chondroitin sulphate 400 mg thrice daily before meals. Period: 127 days
  Other Names: Cosamin DS®; glucosamine hydrochloride and chondroitin sulphate
  Arms: Cosamin DS®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of glucosamine and chondroitin sulfate association in the treatment of patients with osteoarthrosis of the knee.

DETAILED DESCRIPTION:
To assess the efficacy and safety of the association of glucosamine sulphate 500 mg/chondroitin sulphate 400 mg (Eurofarma) in the treatment of osteoarthritis, compared to Cosamin DS® (Nutramax) in same presentation and pharmaceutical form.

Some eligibility criteria:

Osteoarthritis of the knee confirmed by radiological examination; Visual analogue scale (VAS) > 40 mm; Clinical diagnosis of pain and functional limitation

ELIGIBILITY:
Inclusion Criteria:

* Subjects have to read and sign the approved the Informed Consent form prior to any participation in the study.
* Male or female Subjects, aged upper to 40 years.
* Osteoarthritis of the knee confirmed by radiological examination.
* Visual analogue scale (VAS) > 40 mm.
* Kellgren and Lawrence grade 1 to 3.
* Clinical diagnosis of pain and functional limitation.

Exclusion Criteria:

* History of significant trauma or surgery in the affected joint.
* Pregnant women, lactating or not using appropriate contraceptive method.
* History or presence of active rheumatic disease that may be responsible for secondary osteoarthritis.
* Severe inflammation of the joint confirmed by physical examination (excluding also erythrocyte sedimentation <40mm/h and rheumatoid factor <1:40).
* Body mass index > 30.
* Hematologic abnormalities, liver, renal or metabolic functions which undermine the serious participation of the patient (at investigator's criteria).
* Systemic administration and/or intra-articular corticosteroids in the last 3 months.
* Have made use of glucosamine and/or chondroitin.
* Lequesne index of > 12.
* Arthroplasty in the affected joint.
* Use of narcotic analgesics.
* Any condition that, in the opinion of the investigator, renders the patient unable to participate in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Brandão, Phd/MD, Principal Investigator — Centro de Pesquisa Clínica Perdizes; Marise L. Castro, Phd/MD, Principal Investigator — Instituto de Medicina Avancada; Cristiano F. Zerbini, Phd/MD, Principal Investigator — Centro Paulista de Investigacoes Clínicas Ltda.; Jose A. Mendonça, Phd/MD, Principal Investigator — Instituo de Pesquisa Clínica e Assistencia Medica de Campinas
Locations (4):
- Brazil (4):
  - Instituto de Pesquisa Clínica e Assistencia Medica de Campinas, Campinas, São Paulo
  - Centro Paulista de Investigacoes Clinicas Ltda, São Paulo
  - Centro de Pesquisa Clínica Perdizes, São Paulo
  - Instituto de Medicina Avancada, São Paulo

REFERENCES:
- [Derived] Lomonte ABV, Mendonca JA, de Castro Brandao G, Castro ML. Multicenter, randomized, double-blind clinical trial to evaluate efficacy and safety of combined glucosamine sulfate and chondroitin sulfate capsules for treating knee osteoarthritis. Adv Rheumatol. 2018 Dec 5;58(1):41. doi: 10.1186/s42358-018-0041-9. PMID 30657100

RESULTS

PARTICIPANT FLOW:
Groups:
- Glucosamine/Chondroitin Sulphate: Glucosamine hydrochloride 500 mg and chondroitin sulphate 400 mg association (Eurofarma) T.I.D. before each meal
Period: Overall Study
Arm/Group | Cosamin DS® | Glucosamine/Chondroitin Sulphate
Started | 50 | 50
Completed | 44 | 45
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cosamin DS® | Glucosamine/Chondroitin Sulphate | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 28 | 50
  >=65 years | 22 | 17 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.2) | 63.4 (8.3) | 63.7 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 83
  Male | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 44 | 45 | 89

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Efficacy and Safety of the Association of Glucosamine Sulphate 500 mg/Chondroitin Sulphate 400 mg (Eurofarma) in the Treatment of Osteoarthritis, Compared to Cosamin DS® (Nutramax)in Same Presentation and Pharmaceutical Form
Description: To assess the efficacy and safety of the association of glucosamine sulphate 500 mg/chondroitin sulphate 400 mg (Eurofarma) in the treatment of osteoarthritis, compared to Cosamin DS® (Nutramax) in same presentation and pharmaceutical form.
Time Frame: approximately 5 months
Population: In this section the population analyzed was per protocol (PP).
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- Glucosamine/Chondroitin Sulphate: Glucosamine hydrochloride 500 mg and chondroitin sulphate 400 mg association (Eurofarma) T.I.D. before each meal
  Glucosamine sulphate and chondroitin sulphate association: glucosamine sulphate 500 mg and chondroitin sulphate 400 mg association T.I.D. before each meal
Arm/Group | Cosamin DS® | Glucosamine/Chondroitin Sulphate
Number analyzed (Participants) | 41 | 45
percentage of participants | 85.4 [70.1 to 93.4] | 88.9 [75.2 to 95.8]
Statistical Analysis 1: Comparison: Cosamin DS® vs Glucosamine/Chondroitin Sulphate; Test type: Non-Inferiority — Non-inferiority test of Ártico vs Cosamin DS® regarding the decrease of pain scale (VAS) in the PP population (N = 86); p < 0.05, t-test, 1 sided — For numeric variables Test -t student or ANOVA will be used. It will be considered statistically significant P-value less than 0,05

ADVERSE EVENTS:
Groups:
- Cosamin DS®: Glucosamine hydrochloride 500 mg and chondroitin sulphate 400 mg association (Eurofarma) T.I.D. before each meal
- Glucosamine/Chondroitin Sulphate: Glucosamine 500 mg and chondroitin sulphate 400 mg association (Eurofarma) T.I.D. before each meal
Arm/Group | Cosamin DS® | Glucosamine/Chondroitin Sulphate
Serious Adverse Events (participants affected / at risk) | 3/50 | 1/50
Other Adverse Events (participants affected / at risk) | 5/50 | 8/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cosamin DS® (N=50) | Glucosamine/Chondroitin Sulphate (N=50)
Arm fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heart attack (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cosamin DS® (N=50) | Glucosamine/Chondroitin Sulphate (N=50)
headache (General disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 3 (3) | 1 (1)
Nausea (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Worsening Diabetes Mellitus (Endocrine disorders) | 1 (1) | 2 (2)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dyspepsia (Endocrine disorders) | 0 (0) | 1 (1)
Epigastralgia (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No